CLINICAL TRIAL: NCT00979628
Title: Basal Bolus Versus Basal Insulin Regimen for the Treatment of Hospitalized Patients With Type 2 Diabetes Mellitus
Brief Title: Basal Bolus Versus Basal Insulin in Type 2 Diabetes Mellitus (T2DM)
Acronym: Basal-Plus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Guillermo Umpierrez, MD (Other)
Collaborators: Sanofi (Industry); Medical University of South Carolina (Other); Texas A&M University (Other)
Responsible Party: Sponsor-Investigator, Guillermo Umpierrez, MD, Professor of Medicine, Emory University
Organization: Emory University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00020328a
Record Dates: First submitted 2009-09-16; First posted 2009-09-18 (Estimated); Results first posted 2014-04-24 (Estimated); Last update posted 2018-10-10 (Actual); Status verified 2018-09

CONDITIONS: Type 2 Diabetes; Hyperglycemia
Keywords: Type 2 Diabetes; Inpatient Hyperglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hyperglycemia | interventions — Insulin; Insulin Glargine; insulin glulisine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Basal Plus Regimen (Experimental): glargine subcutaneously once daily plus corrective doses of glulisine subcutaneously before meals and bedtime as needed
  Interventions: Drug: Basal Plus
- Basal Bolus (Experimental): glargine subcutaneously once daily plus glulisine subcutaneously before meals (plus corrective doses of glulisine as needed)
  Interventions: Drug: Basal Bolus
- sliding scale regular insulin (SSRI) (Active Comparator): sliding scale regular insulin subcutaneously four-times daily in patients with T2DM admitted to general medicine and surgery wards.
  Interventions: Drug: sliding scale regular insulin (SSRI)

INTERVENTIONS:
Drug: sliding scale regular insulin (SSRI) — four-time daily in patients with T2DM admitted to general medicine and surgery wards.
  Other Names: Novolin R
  Arms: sliding scale regular insulin (SSRI)
Drug: Basal Bolus — glargine once daily plus glulisine before meals (plus corrective doses of glulisine as needed)
  Other Names: Lantus (insulin glargine); Apidra (insulin glulisine)
  Arms: Basal Bolus
Drug: Basal Plus — glargine once daily plus corrective doses of glulisine before meals and bedtime as needed
  Other Names: Lantus (insulin glargine); Apidra (insulin glulisine)
  Arms: Basal Plus Regimen

SUMMARY:
The study is a prospective randomized study comparing safety and effectiveness of a basal-bolus regimen with glargine once daily and glulisine before meals, a basal plus regimen with glargine once daily and supplemental doses of glulisine, and sliding scale regular insulin (SSI) on correction of insulin regimen for the hospital management of medical and surgical patients with type 2 diabetes.

DETAILED DESCRIPTION:
High blood glucose levels in medical and surgery patients with diabetes are associated with increased risk of in-hospital complications and death. Improved glucose control with insulin injections may improve clinical outcome and prevent some of the hospital complications. Numerous studies have shown that high blood glucose increases the risk of wound infection, kidney failure and death. It is not known; however, what is the best insulin regimen in patients who will undergo surgery. The use of repeated injections of regular insulin is commonly used for glucose control in hospitalized patients with diabetes. Recently, the combination of Lantus® and Apidra® insulins has been shown to improve glucose control with lower rate of hypoglycemia (low blood sugar). The investigators' recent preliminary data also indicate that a single daily dose of glargine plus corrective doses of glulisine before meals if needed (Basal Plus) is effective in the management of medical and surgical patients with type 2 diabetes mellitus (T2DM). The average daily blood glucose (BG) levels in patients treated with Basal Plus is equivalent to levels in patients treated with Basal Bolus with glargine once daily plus glulisine before meals (basal bolus regimen). The mean daily BG levels in patients treated with basal plus are lower than those reported in patients treated with sliding scale regular insulin (SSRI). Accordingly, the present study aims to determine which insulin treatment is best for glucose control in hospitalized patients with diabetes admitted to general medicine wards. Glargine, glulisine, and regular insulins are approved for use in the treatment of patients with diabetes by the FDA. A total of 375 subjects with type 2 diabetes will be recruited in this study. The sites for this study are Grady Memorial Hospital, Emory University Hospital, the Atlanta VA Medical Center, Scott & White Memorial Hospital and Clinic, and Medical University of South Carolina.

ELIGIBILITY:
Inclusion Criteria:

* Males or females between the ages of 18 and 75 years admitted to a general medicine or surgical services.
* A known history of type 2 diabetes mellitus > 3 months, receiving either diet alone, oral monotherapy, or with any combination of oral antidiabetic agents (sulfonylureas, meglitinides, metformin, thiazolidinediones, dipeptidyl peptidase (DPP) IV inhibitors).
* Patients admitted for non-cardiac elective or emergency surgery or trauma.
* Subjects must have an admission BG > 140 mg and < 400 mg/dL without laboratory evidence of diabetic ketoacidosis (bicarbonate < 18 milliequivalent /L, potential hydrogen (pH) < 7.30, or positive serum or urinary ketones).

Exclusion Criteria:

* Subjects with increased blood glucose concentration, but without a known history of diabetes (stress hyperglycemia).
* Subjects with a history of diabetic ketoacidosis and hyperosmolar hyperglycemic state, or ketonuria [32].
* Patients with acute critical or surgical illness admitted to the ICU or expected to require admission to the ICU.
* Patients admitted for coronary artery bypass graft (CABG) or patients receiving continuous insulin infusion.
* Patients with clinically relevant hepatic disease (diagnosed liver cirrhosis and portal hypertension), corticosteroid therapy, or impaired renal function (creatinine ≥ 3.0 mg/dl).
* Mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study.
* Female subjects are pregnant or breast feeding at time of enrollment into the study.
* Patients with recognized or suspected endocrine disorders associated with increased insulin resistance, acromegaly, or hyperthyroidism.
* Female subjects are pregnant or breast feeding at time of enrollment into the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 375 (Actual)
Dates: Start 2010-01; Primary Completion 2012-03 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Umpierrez, MD, Principal Investigator — Emory SOM
Locations (5):
- United States (5):
  - Grady Memorial Hospital, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Atlanta VA Medical Center, Decatur, Georgia
  - Medical University of South Carolina, Charleston, South Carolina
  - Scott & White Memorial Hospital and Clinic, Temple, Texas

REFERENCES:
- [Result] Umpierrez GE, Smiley D, Hermayer K, Khan A, Olson DE, Newton C, Jacobs S, Rizzo M, Peng L, Reyes D, Pinzon I, Fereira ME, Hunt V, Gore A, Toyoshima MT, Fonseca VA. Randomized study comparing a Basal-bolus with a basal plus correction insulin regimen for the hospital management of medical and surgical patients with type 2 diabetes: basal plus trial. Diabetes Care. 2013 Aug;36(8):2169-74. doi: 10.2337/dc12-1988. Epub 2013 Feb 22. PMID 23435159
- [Derived] Umpierrez GE, Reyes D, Smiley D, Hermayer K, Khan A, Olson DE, Pasquel F, Jacobs S, Newton C, Peng L, Fonseca V. Hospital discharge algorithm based on admission HbA1c for the management of patients with type 2 diabetes. Diabetes Care. 2014 Nov;37(11):2934-9. doi: 10.2337/dc14-0479. Epub 2014 Aug 28. PMID 25168125

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 375 subjects were enrolled in the study from January 2010 to June 2012. The study is conducted in 3 states and patients were enrolled from 3 hospitals in state of Georgia; 1 hospitals in south Carolina and 1 hospitals in Texas.
Pre-assignment Details: 24 subjects that were consented were withdrawn from the study and not included in analysis because they meet exclusion criteria like transferring to ICU; receiving treatment < 24 hrs and for receiving steroids
Groups:
- Basal Bolus: glargine once daily plus glulisine before meals (plus corrective doses of glulisine as needed)
  Basal Bolus : glargine once daily plus glulisine before meals (plus corrective doses of glulisine as needed)
- Basal Plus Regimen: glargine once daily plus corrective doses of glulisine before meals and bedtime as needed
  Basal Plus : glargine once daily plus corrective doses of glulisine before meals and bedtime as needed
- Sliding Scale Regular Insulin (SSRI): four-time daily in patients with T2DM admitted to general medicine and surgery wards.
  sliding scale regular insulin (SSRI) : four-time daily in patients with T2DM admitted to general medicine and surgery wards.
Period: Overall Study
Arm/Group | Basal Bolus | Basal Plus Regimen | Sliding Scale Regular Insulin (SSRI)
Started | 153 | 142 | 80
Completed | 144 | 133 | 74
Not Completed | 9 | 9 | 6
Not completed — received regimen < 24 hours | 7 | 6 | 5
Not completed — received steroids | 1 | 1 | 0
Not completed — transferred to ICU | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Basal Bolus: glargine once daily plus glulisine before meals (plus corrective doses of glulisine as needed)
  Basal Bolus : glargine once daily plus glulisine before meals subcut at an initial dose of 0.3-0.5 units/kg/day (plus corrective doses of glulisine as needed)
- Basal Plus Regimen: glargine once daily plus corrective doses of glulisine before meals and bedtime as needed
  Basal Plus : glargine once daily subcut at an initial dose of 0.15-0.25 units/kg/day plus corrective doses of glulisine subcut before meals and bedtime as needed
- Sliding Scale Regular Insulin (SSRI): four-time daily in patients with T2DM admitted to general medicine and surgery wards.
  sliding scale regular insulin (SSRI) given subcut four-times daily before meals and at bedtime
- Total: Total of all reporting groups
Arm/Group | Basal Bolus | Basal Plus Regimen | Sliding Scale Regular Insulin (SSRI) | Total
Number analyzed (Participants) | 153 | 142 | 80 | 375
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.7 (11) | 58.6 (13) | 58.7 (12) | 58.6 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 65 | 33 | 160
  Male | 91 | 77 | 47 | 215

OUTCOME MEASURES:

1. Primary Outcome: Mean Blood Glucose Levels (Measured in mg/dL) at Randomization Are Compared to Mean Blood Glucose Levels After First Day of Treatment Among Subjects Treated With Basal Plus, Basal -Bolus and SSRI Treatments
Description: The primary outcome is to determine the effective glycemic control among the subjects that received Basal Plus (glargine once daily plus corrective doses of glulisine before meals and bedtime as needed), Basal Bolus approach of glargine once daily plus corrective doses of glulisine before meals and Sliding Scale Regular Insulin (SSRI). Glycemic control is measured by mean blood glucose(BG) levels in mg/dL after first day of treatment and are compared to mean BG levels at randomization among subjects treated with Basal Plus, Basal -bolus and SSRI treatments. The optimal glycemic control is achieved when BG levels are between 70 mg/dL -140 mg/dL. The BG levels levels below 70 mg/dL are regarded as hypoglycemic events. The BG levels levels above 140 mg/dl are considered elevated and Hyperglycemia defined as a fasting BG >126 mg/dl or random BG >200 mg/dl on two or more occasions).
Time Frame: Randomization and 24 hrs after treatment
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Basal Plus Regimen: glargine once daily plus corrective doses of glulisine before meals and bedtime as needed
  Basal Plus: glargine once daily plus corrective doses of glulisine before meals and bedtime as needed
- Sliding Scale Regular Insulin (SSRI): four-time daily in patients with type 2 diabetes mellitus (T2DM) admitted to general medicine and surgery wards.
  sliding scale regular insulin (SSRI): four-time daily in patients with T2DM admitted to general medicine and surgery wards.
Arm/Group | Basal Plus Regimen | Basal Bolus | Sliding Scale Regular Insulin (SSRI)
Number analyzed (Participants) | 133 | 144 | 74
mg/dL
  Randomization | 194 (45) | 200 (49) | 187 (43)
  After first day of therapy | 163 (37) | 156 (36) | 172 (41)

2. Secondary Outcome: Number of Patients With Hypoglycemia Events (Blood Glucose Levels < 70 mg/dL) During Their Hospital Stay That Are Treated With Basal Plus, Basal-bolus and SSRI Treatments
Description: Effective Glycemic control is also assessed by number of hypoglycemia events among the patients treated with Basal plus, basal-bolus and SSRI treatments. Hypoglycemia event is defined as blood glucose levels <70 mg/dL. Number of patients with hypoglycemia episodes that are treated with Basal plus, basal-bolus and SSRI treatment regimens during their hospital stay are examined and compared.
Time Frame: During hospital stay, up to 12 days
Measure: Number; unit: participants
Arm/Group | Basal Bolus | Basal Plus Regimen | Sliding Scale Regular Insulin (SSRI)
Number analyzed (Participants) | 144 | 133 | 74
participants | 23 | 17 | 2

ADVERSE EVENTS:
Time Frame: The time frame for the study is the duration of hospital stay of the patients. Among the study patients the mean (standard deviation) hospital stay for Basal bolus patients was 5.9 (5) days; Basal plus patients was 6(6) days; SSRI patients was 5.5(5) days.
Description: Subjects were followed daily by the investigators for complications and mortality. But the study end points on adverse events are related to blood glucose (BG) levels. Hypoglycemia is defined as BG levels of < 70 mg/dL. Severe hypoglycemia is defined as blood glucose levels of < 40 mg/dL. Inpatient hyperglycemia defined as a fasting BG >126 mg/dl or random BG >200 mg/dl on two or more occasions.
Arm/Group | Basal Plus Regimen | Basal Bolus | Sliding Scale Regular Insulin (SSRI)
All-Cause Mortality (participants affected / at risk) | 3/133 | 0/144 | 0/74
Serious Adverse Events (participants affected / at risk) | 18/133 | 22/144 | 7/74
Other Adverse Events (participants affected / at risk) | 16/133 | 13/144 | 3/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Basal Plus Regimen (N=133) | Basal Bolus (N=144) | Sliding Scale Regular Insulin (SSRI) (N=74)
Severe hypoglycemia (Metabolism and nutrition disorders) | 1 | 1 | 0 — blood glucose < 40 mg/dl
wound infections (Infections and infestations) | 3 | 1 | 1
pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Acute Renal Failure (Renal and urinary disorders) | 8 | 9 | 3
Bacteremia (Infections and infestations) | 4 | 7 | 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Basal Plus Regimen (N=133) | Basal Bolus (N=144) | Sliding Scale Regular Insulin (SSRI) (N=74)
Hypoglycemia (Metabolism and nutrition disorders) | 16 | 13 | 3 — blood glucose < 70 mg/dl

LIMITATIONS AND CAVEATS:
- The study excluded patients admitted to the ICU, those with clinically relevant hepatic disease or with serum creatinine >3.0 mg/dL, patients with severe hyperglycemia, and those receiving a total dose of insulin >0.4 units/kg/day before admission.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No